CLINICAL TRIAL: NCT01125839
Title: Clinical Features, Microbiological-, Radiological Characteristics, and Differential Diagnosis of Vertebral Osteomyelitis
Brief Title: Characterization and Differential Diagnosis of Vertebral Osteomyelitis
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang-Ho Choi, Doctor, Asan Medical Center
Other Study IDs: AVOMS
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2013-09

CONDITIONS: Vertebral Osteomyelitis
Keywords: osteomyelitis; 16S rRNA; spine; Magnetic resonance imaging
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CT guided biopsy specimen
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Spondylitis: Patients who checked spine MRI for back pain

SUMMARY:
Vertebral osteomyelitis is a uncommon disease that can lead to neurologic deficits if not diagnosed in time. The etiologies of vertebral osteomyelitis include pyogenic bacteria, M. tuberculosis, Brucella species, and fungus. The aim of this study is to describe the clinical features and microbiological/radiological characteristics of patients with vertebral osteomyelitis, and investigate the useful tips for the differential diagnosis of vertebral osteomyelitis.

DETAILED DESCRIPTION:
Besides description of characteristics of patients with vertebral osteomyelitis, we also will investigate the usefulness of 16S rRNA gene sequence analysis of biopsy specimen. MRI findings during the antibiotic treatment will be monitored and compared for the differential diagnosis of meningitis.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms or signs consistent with spinal column infection
* MRI findings suggestive of infection
* Antibiotic treatment for vertebral myelitis

Exclusion Criteria:

* Patients already treated more than 2 weeks for osteomyelitis in transferring hospital

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that have MRI findings sugggestive of vertebral osteomyelitis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Identification of etiology of vertebral osteomyelitis | within 6 weeks after the diagnosis of vertebral osteomyelitis

SECONDARY OUTCOMES:
Unfavorable outcomes (death or permanent neurologic deficit) | within 6 months after the diagnosis of vertebral osteomyelitis

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Ho Choi, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea